CLINICAL TRIAL: NCT04438707
Title: Pilates Method and Therapeutic Exercise in Children That Play String Instruments: Pilot Study
Brief Title: Pilates Method and Therapeutic Exercise in Children That Play String Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEUSP
Record Dates: First submitted 2020-06-01; First posted 2020-06-19 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-06

CONDITIONS: Postural Kyphosis; Postural Lordosis; Postural Low Back Pain
Keywords: Pilates; Therapeutic Exercise; Children; String instruments; Vertebral column
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Pilot study designed by a randomized controlled trial in two parallel intervention groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: Pilates Method combined with Therapeutic exercice.
- Control group (Active Comparator)
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Pilates Method combined with Therapeutic exercice. — Children must perform specific exercices in this combined method with the pilates principes (for back) during 50 min (1 day per week) for 4 weeks.
  Arms: Experimental group
Other: Therapeutic exercise — Children must perform specific exercices without the pilates principes (for back) during 50 min (1 day per week) for 4 weeks.
  Arms: Control group

SUMMARY:
Introduction: An inappropriate posture in children for a while kept playing some instrument of the group of the rubbed string, can cause pain and alterations of the spine, as it continues to consolidate.

Objective: To study the benefits acquired during the application of the Pilates Method combined with therapeutic exercise against the Therapeutic Exercise to reduce alterations of the vertebral rachis in children from 10 to 14 years old who play instruments of rubbed strings.

DETAILED DESCRIPTION:
Material and methods: A pilot study designed by a randomized controlled trial in two parallel intervention groups was carried out; 9 children performed the combination of the Pilates Method and Therapeutic Exercise (experimental) and 7 children performed the Therapeutic Exercise (control). At the beginning and at the end of the study, pain measurements have been made through the Visual Analogue Scale (EVA), and the Kinovea programme for the alignment of shoulder, scapula and hip postures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with typical development and ages between 10 and 14 years old.
* Subjects who play the violin, viola, cello or double bass. Subjects who have learned to play the violin, viola, cello or double bass in this school year or up to a maximum of four previous years, eligible to receive Pilates classes.
* Subjects with cognitive ability to understand simple orders.
* Subjects who are enrolled this year in Orchestrated Neighborhoods.

Exclusion Criteria:

* Subjects whose ages are not between 10 and 14 years of age.
* Subjects who do not play the violin, viola, cello, or double bass.Subjects who have more than four school years playing the violin, viola, cello or double bass.
* Subjects who do not have cognitive capacity to understand simple orders.
* Subjects who are not registered this year in Orchestrated Neighborhoods.
* Subjects who do not complete the four sessions of Therapeutic Exercise + Pilates or Therapeutic Exercise.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
SVA | 4 weeks
  to assess the pain in children. The child must choose a number (0-10) depending of the pain intensity.

SECONDARY OUTCOMES:
Kinovea tool | 4 weeks
  to assess the alignement in shoulders, hips. It meusered in degrees of movement to observe the amplitud in the movemente and the simetry of joints. It is used a software to analyse the information and obtain the posture in the child.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Poncela, Therapyst, Principal Investigator — CEU San Pablo University
Locations (1):
- Carolina Poncela, Santa Cruz de Tenerife, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will show the study protocol, de statistical resulst done with SPSS and the informed consent form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the study is finished and all the data are analized by SPSS. It will be available for 6 months.